CLINICAL TRIAL: NCT00199329
Title: Antiemetic Effect of the Addition of Ondansetron to the Morphine Solution in Patient-Controlled Analgesia (PCA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: I48027
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2007-10

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: ondansetron; PCA
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: ondansetron adding in PCA

SUMMARY:
PCA morphine always introduces nausea and vomiting during the postoperative period. Ondansetron can reduce PONV (postoperative nausea vomiting). We, the researchers at Khon Kaen University, are trying to add ondansetron in PCA morphine. Patients receive a small dose of ondansetron when they request morphine.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15-60 years old

Exclusion Criteria:

* History of motion sickness, smoking

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 160 (Actual)
Dates: Start 2005-01

PRIMARY OUTCOMES:
PONV | 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Polpun Boonmak, MD, Study Director — lecturer in Khon Kaen University
Locations (1):
- Khon Kaen university, Srinagarind Hospital, Muang, Changwat Khon Kaen, Thailand